CLINICAL TRIAL: NCT02680041
Title: The Impact of 18F Fluciclovine (FACBC) PET/CT (Positron Emission Computed Tomography) on Management of Patients With Rising PSA (Prostate-specific Antigen) After Initial Prostate Cancer Treatment
Brief Title: 18F Fluciclovine (FACBC) PET/CT in Patients With Rising PSA After Initial Prostate Cancer Treatment
Acronym: LOCATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Blue Earth Diagnostics (Industry)
Collaborators: American College of Radiology (Other); IND 2 Results LLC (Industry); Syne Qua Non Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BED003
Record Dates: First submitted 2016-01-15; First posted 2016-02-11 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-fluciclovine PET CT (Experimental): Single intravenous administration of 18F-fluciclovine PET CT.
  Interventions: Drug: 18F-fluciclovine PET CT

INTERVENTIONS:
Drug: 18F-fluciclovine PET CT — Subjects will undergo a fluciclovine F18 PET/CT scan in addition to standard of care monitoring. The results of this scan may influence further treatment
  Other Names: FACBC

SUMMARY:
This prospective study will enroll up to 330 men with PSA-persistent or PSA-recurrent prostate cancer after curative-intent primary therapy and negative or equivocal findings on standard-of-care imaging. Consenting participants will be imaged with 18F-fluciclovine PET/CT. Site clinicians will manage study subjects per standard practices and will document any change in treatment based on review of 18F-fluciclovine PET/CT findings. All participants will be followed for up to 6 months, with clinical data collected for this study. An interdisciplinary panel will provide expert guidance to local readers on request. The final reporting of the PET/CT scan will be a single report by the local reader following any such discussion.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed adenocarcinoma of the prostate post curative-intent local treatment (radical prostatectomy, local radiotherapy, brachytherapy).
* Suspicion of recurrent prostate carcinoma after previous presumed definitive therapy for organ confined disease defined as :
* Post prostatectomy: Detectable or rising PSA level that is >0.2 ng/mL with a second confirmatory level of >0.2 ng/mL
* Post non-prostatectomy: PSA rise ≥ 2ng/mL over nadir
* Negative or equivocal findings on standard-of-care imaging for restaging of disease in the previous 60 days consisting of: Whole-body 99mTc bone scintigraphy or NaF PET-CT; and either CT or MRI of the pelvis (or the abdomen and pelvis).
* Being considered for salvage therapy
* Any non-surgical local treatment such as previous cryotherapy, external beam radiation, or HiFU (Ultrasound) must have occurred at least 1 year in the past.
* Previous brachytherapy treatment will have occurred at least 2 years in the past
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Ongoing treatment with any systemic therapy intended for the treatment of prostate cancer (e.g., antiandrogen or LHRH agonist or antagonist)
* Androgen deprivation therapy (ADT) in the past 3 months
* History of bilateral orchidectomy
* Inability to tolerate 18F-fluciclovine PET/CT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Umar Mahmood, MD, PhD, Study Chair — Harvard Medical School (HMS and HSDM); Peter Gardiner, MB ChB, MRCP, FFPM, Study Director — Blue Earth Diagnostics
Locations (17):
- United States (17):
  - City of Hope National Medical Center, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Tower Urology, Los Angeles, California
  - Genesis Research, LLC, San Diego, California
  - University of Florida, Jacksonville, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Roudebush VA Medical Center, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - Coastal Urology Associates, Brick, New Jersey
  - Manhattan Medical Research, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Urologic Consultants of SE Pennsylvania, Bala-Cynwyd, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andriole GL, Scarsbrook AF, Savir-Baruch B; LOCATE/FALCON Study Groups. Impact of 18F-fluciclovine PET/CT on plans for androgen deprivation therapy in patients with biochemical recurrence of prostate cancer: data analysis from two prospective clinical trials. Urol Oncol. 2023 Jun;41(6):293.e1-293.e7. doi: 10.1016/j.urolonc.2023.04.004. Epub 2023 Apr 29. PMID 37121865
- [Derived] Savir-Baruch B, Lovrec P, Solanki AA, Adams WH, Yonover PM, Gupta G, Schuster DM. Fluorine-18-Labeled Fluciclovine PET/CT in Clinical Practice: Factors Affecting the Rate of Detection of Recurrent Prostate Cancer. AJR Am J Roentgenol. 2019 Oct;213(4):851-858. doi: 10.2214/AJR.19.21153. Epub 2019 Jun 19. PMID 31216198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 01 June 2016 (first patient, screening visit) and 01 November 2017 (last patient, last contact) at 17 sites in the USA. Overall 17 sites were initiated, of which 15 sites enrolled patients.
Period: Overall Study
Arm/Group | 18F-fluciclovine PET CT
Started | 221
Received 18F-fluciclovine | 213
Completed | 211
Not Completed | 10
Not completed — Withdrawal prior to 18F-fluciclovine PET | 8
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- 18F-fluciclovine PET CT: Single intravenous administration of 18F-fluciclovine PET/CT.
Arm/Group | 18F-fluciclovine PET CT
Number analyzed (Participants) | 213
Age, Continuous [Median (Full Range); unit: years] | 67.0 [46 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 202
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 17
  White | 188
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 213

OUTCOME MEASURES:

1. Primary Outcome: The Fraction of Patients for Whom 18F-fluciclovine PET/CT Alters Patient Planned Treatment Through Detection of Disease.
Description: The change of management will be based on referring physician questionnaires completed pre- and post- 18F-fluciclovine PET/CT
Time Frame: 2-22 days post PET CT
Population: For the primary analysis population, of the 213 patients included in the EAS, 122 patients with a positive 18F-fluciclovine scan and 91 patients with a negative 18F-fluciclovine scan had a pre 18F-fluciclovine PET/CT treatment management plan.
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-fluciclovine PET CT
Number analyzed (Participants) | 213
Participants
  Overall Evaluable Analysis Set: Patients with Revised Management Plan | 126
  Overall Evaluable Analysis Set: No Revision to Management Plan | 87
  Positive 18F-fluciclovine Scan: number analyzed (Participants) | 122
  Positive 18F-fluciclovine Scan: Patients with Revised Management Plan | 88
  Positive 18F-fluciclovine Scan: No Revision to Management Plan | 34
  Negative 18F-fluciclovine Scan: number analyzed (Participants) | 91
  Negative 18F-fluciclovine Scan: Patients with Revised Management Plan | 38
  Negative 18F-fluciclovine Scan: No Revision to Management Plan | 53

2. Secondary Outcome: The Fraction of Patients for Whom 18F-fluciclovine PET/CT Alters Patient Actual Treatment
Description: The change of management will be based on referring physician questionnaires completed pre- 18F-fluciclovine PET/CT and changes reported at 6 month follow-up.
  Investigators were instructed to assess any clinically significant change from the revised management plan.
Time Frame: 6 months
Population: 211 participants completed the study (actual treatment assessed at study completion).
  Results also presented by 18F-fluciclovine PET CT results.
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-fluciclovine PET CT
Number analyzed (Participants) | 211
Participants
  Overall: Change from the revised management plan | 80
  Overall: No change from the revised management plan | 131
  Positive 18F fluciclovine Scan: number analyzed (Participants) | 121
  Positive 18F fluciclovine Scan: Change from the revised management plan | 47
  Positive 18F fluciclovine Scan: No change from the revised management plan | 74
  Negative 18F fluciclovine Scan: number analyzed (Participants) | 90
  Negative 18F fluciclovine Scan: Change from the revised management plan | 33
  Negative 18F fluciclovine Scan: No change from the revised management plan | 57

3. Secondary Outcome: The Rate of Detection of Any Disease Site by 18F-fluciclovine PET/CT in the Study Population
Description: The percentage of subjects who have disease detectable by 18F-fluciclovine PET/CT
Time Frame: 1 week
Population: Results presented for Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-fluciclovine PET CT
Number analyzed (Participants) | 213
Participants | 122

4. Secondary Outcome: The Rate of Detection of Disease in 1) Prostate and Prostate Bed and 2) Extra-prostatic Regions With 18F-fluciclovine PET/CT in the Study Population
Description: The percentage of subjects who have disease detectable by 18F-fluciclovine PET/CT 1) in the pelvis and 2) distally
Time Frame: 1 week
Population: Participants may have lesions detected in both regions (prostate/prostate bed and extra-prostatic).
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-fluciclovine PET CT
Number analyzed (Participants) | 213
Participants
  Prostate or Prostate Bed | 64
  Extra-prostatic | 80

5. Secondary Outcome: The Positive Predictive Value (PPV) of 18F-fluciclovine PET/CT for Regional Disease Compared to Biopsy in Those Patients Who Undergo Biopsy or in Case of Bony Disease a Correlation With MRI or Biopsy
Description: Based on the ratio of positive findings in the pelvis on 18F-fluciclovine PET/CT which are confirmed by histological examination of tissue or MRI
Time Frame: 6 months
Population: Only scans graded as positive or negative by the adjudication panel were included in these calculations.
Measure: Number (95% Confidence Interval); unit: Percentage of scans
Arm/Group | 18F-fluciclovine PET CT
Number analyzed (Participants) | 45
Percentage of scans | 100 [92.1 to 100.0]

6. Secondary Outcome: The PPV of 18F-fluciclovine PET/CT for Distant Disease Compared to Biopsy in Those Patients Who Undergo a Biopsy or in Case of Bony Disease a Correlation With MRI or Biopsy
Description: Based on the ratio of positive findings outside the pelvis on 18F-fluciclovine PET/CT which are confirmed by histological examination of tissue or MRI
Time Frame: 6 months
Population: Only scans graded as positive or negative by the adjudication panel were included in these calculations.
Measure: Number (95% Confidence Interval); unit: Percentage of scans
Arm/Group | 18F-fluciclovine PET CT
Number analyzed (Participants) | 37
Percentage of scans | 100 [90.5 to 100.0]

ADVERSE EVENTS:
Time Frame: As specified in the Statistical Analysis Plan, results are presented as only those treatment-emergent adverse events which occurred up to 42 days after the 18F fluciclovine administration.
Arm/Group | 18F-fluciclovine PET CT
All-Cause Mortality (participants affected / at risk) | 0/213
Serious Adverse Events (participants affected / at risk) | 0/213
Other Adverse Events (participants affected / at risk) | 44/213
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 18F-fluciclovine PET CT (N=213)
Diarrhoea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 2
Oedema peripheral (General disorders) | 2
Headache (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Urinary Tract Infection (Infections and infestations) | 2
Hot flush (Vascular disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Stress urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Excercise tolerance decreased (General disorders) | 1
Fatigue (General disorders) | 1
Feeling cold (General disorders) | 1
Injection site extravasation (General disorders) | 1
Injection site pain (General disorders) | 1
Pyrexia (General disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intervertrabral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Emotional disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Listless (Psychiatric disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal abscess (Infections and infestations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatine increased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Carbon dioxide decreased (Investigations) | 1
Waist circumference increased (Investigations) | 1
Breast tenderness (Reproductive system and breast disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 1
Scrotal irritation (Reproductive system and breast disorders) | 1
Atrial fibrilation (Cardiac disorders) | 1
Hyperchloreamia (Metabolism and nutrition disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor Investigator will submit for publication or public disclosure any publication or disclosure based on the results of the Study until after the first to occur of (a) publication of the Multi-Center Clinical Trial results; (b) notification by Sponsor that the Multi-Center Clinical Trial submission is no longer planned; or (c) the eighteen (18) month anniversary of the completion or early termination of the Multi-Center Clinical Trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT02680041/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT02680041/SAP_001.pdf